CLINICAL TRIAL: NCT02558725
Title: Iron Supplementation During Pregnancy - One Versus Two Ferrous Sulfate Capsules for Iron Deficient Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Principal Investigator, maslovitz sharon, Dr, Assuta Hospital Systems
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015057
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Pregnancy Complications, Hematologic
MeSH Terms: conditions — Pregnancy Complications, Hematologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- one capsule of iron supplement (No Intervention): instructed to take one capsule at least 2 hours after consumption of dairy products
- two capsules of iron supplement (Active Comparator): instructed to take two capsules of Aktiferrin F at least 2 hours after consumption of dairy products
  Interventions: Drug: two capsules of aktiferrin F

INTERVENTIONS:
Drug: two capsules of aktiferrin F — two capsules of Aktiferrin F or Foliferrin
  Other Names: Foliferrin
  Arms: two capsules of iron supplement

SUMMARY:
Since normal pregnancies are associated with dilutional anemia, due to a greater increase in plasma volume with a smaller increase in RBC mass, it is important to properly diagnose IDA according to the levels of serum ferritin. Previous studies examining the optimal iron dose have shown that adjustment of iron supplementation according to serum ferritin levels in early pregnancy could be beneficial. Nonetheless, there is no consensus regarding the appropriate dose of iron during pregnancy, its dose-response curve and its effect on serum ferritin levels.

In this trial the investigators sought to assess the efficacy of doubling the daily iron supplement dose in pregnant women with IDA.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled trial performed at a women's health center from April 2015 . All participants had a complete blood count performed during their initial visit to the clinic during the first trimester of pregnancy. IDA was defined as a hemoglobin concentration <10.5 g/dL and ferritin levels < 15 ng/ml.

Inclusion criteria were healthy pregnant women ages 18-42 with a singleton gestation and a diagnosis of IDA between 16-19 weeks. The investigators included only women with full access to medical computerized files. Exclusion criteria were: multiple pregnancies, hyperemesis gravidarum continuing past 20 weeks of gestation, Thalassemia, abnormal blood smears, vitamin D deficiency, mal-absorption disorders (inflammable bowel diseases; Crohn's, Ulcerative Colitis) and chronic diseases associated with anemia (i.e SLE). Vitamin B12 and blood smears were performed at the time of allocation. Additional inclusion criteria applied after allocation were: deterioration in hemoglobin levels mandating IV iron administration, more than 3 capsules missed at the 2 weeks check-up, diarrhea lasting more than 5 days, vomiting lasting more than 5 days less than 2 hours after supplement , administration of blood products during pregnancy, any use of multi-vitamin supplements containing iron, hospitalization periods greater than two weeks and a time period shorter than 15 weeks from allocation to delivery.

All participants diagnosed with IDA fulfilling the inclusion criteria were randomized by "Randomizer" (http://www.randomizer.org) to receive either one or two capsules of aktiferrin F (containing DL-Serine 129 mg; Iron (Ferrous Sulfate) 34 mg; Folic Acid 0.5 mg) or Foliferrin (containing DL-Serine 120 mg; Iron (Ferrous Sulfate) 34 mg; Folic Acid 0.5 mg). No cross-over was permitted between groups.

Participants were instructed to take one capsule at least 2 hours after consumption of dairy products or two capsules 12 hours apart at least 2 hours after consumption of dairy products. Validation of compliance to medical regimens was performed by a count of empty pill packages every two weeks during regular check-ups. All participants were monitored for weight, BP and urine dipstick measurements every 2-3 weeks until 34 weeks. Episodes of vomiting, constipation and diarrhea were recorded. Constipation was defined as fewer than three bowel movements a week or bowel movements consisting of hard, dry and small stool, making it painful or difficult to pass. Fetal BPP and estimated weight were performed every 2-3 weeks until 34 weeks of gestation. Fetal monitor was performed every two weeks from 34 weeks of gestation.

Laboratory follow up was performed by measurements of ferritin and hemoglobin levels at fixed time intervals during gestation: 15-20 weeks, 24 weeks, 35 weeks and also 6 weeks post-partum. All lab studies were performed in a single central laboratory.

The data extracted included demographic data (age, parity, chronic disease, weight and BMI at allocation and weight gain during the study period), obstetrical complications (GDM, preeclampsia, IUGR, preterm labor, preterm delivery, IUFD and blood product transfusion) and non obstetrical complications (diarrhea, thrombocytopenia, gastroenteritis, appendicitis, hypo/hyperthyroidism, pre-gestational diabetes) and newborn outcome (birth-weight and Apgar score and immediate post-partum complications). Any gastrointestinal symptoms, obstetrical complications or hospital admissions were reported in real time to the PI

ELIGIBILITY:
Inclusion Criteria:

1. Healthy pregnant women ages 18-42
2. A diagnosis of iron deficiency anemia (defined as a hemoglobin concentration <10.5 g/dL and ferritin levels < 15 ng/ml) between 16-19 weeks
3. Full access to medical computerized files.

Exclusion Criteria:

1. Hyperemesis gravidarum continuing past 20 weeks of gestation
2. Thalassemia
3. Abnormal blood smears
4. Vitamin D deficiency
5. Mal-absorption disorders (inflammable bowel diseases; Crohn's, Ulcerative Colitis)
6. Chronic diseases associated with anemia (i.e SLE).
7. Deterioration in hemoglobin levels mandating IV iron administration
8. More than 3 capsules missed at the 2 weeks check-up
9. diarrhea lasting more than 5 days
10. Vomiting lasting more than 5 days less than 2 hours after supplement ingestion
11. Administration of blood products during pregnancy
12. Use of multi-vitamin supplements containing iron
13. Hospitalization periods greater than two weeks
14. A time period shorter than 15 weeks from allocation to delivery -

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
mean hemoglobin level | at 35 weeks gestation

SECONDARY OUTCOMES:
mean ferritin level | at 35 weeks
mean hemoglobin level | at 6 weeks post-partum
incidence of constipation | every 2 weeks from 20th week to 40th week
birth-weights | at delivery
mean ferritin level | 6 weeks after delivery
the incidence of preterm birth rate (<37 weeks) | at delievery
NICU admission rate | at 1 week after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Maslovitz, Dr, Principal Investigator — Maccabi Healthcare Services, Israel
Locations (1):
- Assuta Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Shinar S, Skornick-Rapaport A, Maslovitz S. Iron supplementation in singleton pregnancy: Is there a benefit to doubling the dose of elemental iron in iron-deficient pregnant women? a randomized controlled trial. J Perinatol. 2017 Jul;37(7):782-786. doi: 10.1038/jp.2017.43. Epub 2017 Apr 6. PMID 28383533